CLINICAL TRIAL: NCT06484387
Title: Study of Multimodal Intra- and Interpersonal Synchronizations in Social Interaction in Individuals with a Diagnosis of Schizophrenia.
Brief Title: Study of Intra- and Interpersonal Multimodal Synchronizations in a Social Interaction in Individuals with a Diagnosis of Schizophrenia.
Acronym: ENHANCER1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Euromov Digital Health in Motion (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: RECHMPL22_0408
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Schizophrenia
Keywords: social interaction; interpersonal synchronization
MeSH Terms: conditions — Schizophrenia | interventions — Drug Interactions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dyad schizophrenia and interacting partner (Experimental): social interaction between an individual with a diagnosis of schizophrenia and his interacting partner
  Interventions: Behavioral: Social interaction
- dyad healthy subject and interacting partner (Experimental): social interaction between a healthy subject and his interacting partner
  Interventions: Behavioral: Social interaction

INTERVENTIONS:
Behavioral: Social interaction — Participants are required to speak to one another. Participants are given various topics of conversation.

SUMMARY:
The aim of this study is to precisely identify deficits in intra- and interpersonal multimodal synchronizations during social interaction in individuals with schizophrenia (ISZ). During a social interaction, individuals use both visual and auditory channels to construct their discourse. The auditory channel encompasses the semantics and prosody of the speech, while the visual channel describes the entirety of non-verbal gestures (e.g., facial expressions, body movements). Prosody and non-verbal gestures are essential elements for the speaker. By accompanying speech, they contribute to the planning and conceptualization of the utterance and enhance its communicative power. For the listener, prosody and non-verbal gestures are also used to provide sensory feedback to the speaker.

Several studies have shown the existence of intrapersonal and interpersonal synchronizations of prosody and non-verbal gestures during interaction. These synchronizations are associated with numerous social benefits (e.g., increased mutual appreciation and quality of interaction). However, certain mental disorders, such as schizophrenia, exhibit deficits in non-verbal behaviors that can impair these synchronizations and the associated social benefits. We hypothetized that interaction with individuals with a daignosis of schizophrenia will be associated with deficits in intra and interpersonal synchronization.

DETAILED DESCRIPTION:
This study includes a pre-inclusion interview followed by a visit to the university hospital (CHU) lasting about 2 hours (including a break). During the visit, the patient participates in an experimental protocol consisting of two parts. In the first part, the patient will be paired with an interaction partner, and the two participants will engage in four distinct conversational tasks, including getting to know each other, free discussions, structured dialogues, and emotional interactions. In the second part, the participants will answer several questionnaires and perform neuropsychological tests in collaboration with an experimenter

ELIGIBILITY:
Individuals with a diagnosis of schizophrenia :

Inclusion Criteria:

* diagnosis of schizophrenia according to the DSM-V
* being able to read, speak and understand french
* giving eclaired consent

Exclusion Criteria:

* history of head trauma
* history of neurological conditions (epilespsy, multiple sclerosis, parkinson's disease, amyotrophic lateral sclerosis, huntington's disease, stroke)
* substance use
* pregnant women

Healthy controls :

Inclusion Criteria:

* being able to read, speak and understand french
* giving eclaired consent

Exclusion Criteria:

* diagnosis of psychosis
* history of head trauma
* history of neurological conditions (epilespsy, multiple sclerosis, parkinson's disease, amyotrophic lateral sclerosis, huntington's disease, stroke)
* substance use
* pregnant women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2025-11-08 (Estimated); Study Completion 2025-11-08 (Estimated)

PRIMARY OUTCOMES:
interpersonal synchronization | 4x6 minutes
  synchronization between body movements of two interacting partners
intrapersonal synchronization | 4x6 minutes
  synchronization between voice and body movements of one individual

SECONDARY OUTCOMES:
correlation between primary outcomes and individuals with schizophrenia medications | 4x6 minutes
correlation between synchronization and willingness to continue the interaction | 4x6 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No